CLINICAL TRIAL: NCT03205384
Title: Analysis of Morbimortality and Functional Status in Older Patients(>65 Years Old) Undergoing Urgent Abdominal Surgery Using CRISTAL Score Modify
Brief Title: Morbimortality in Older Patients Undergoing Urgent Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: Hospital of Navarra (Other)
Responsible Party: Principal Investigator, Ines Eguaras, Principal investigator, Hospital of Navarra
Other Study IDs: CHN
Record Dates: First submitted 2017-02-22; First posted 2017-07-02 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Surgery--Complications
Keywords: Urgent abdominal surgery. Quality of life, functional status, frailty, nutritional status
MeSH Terms: conditions — Frailty | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- surgical management: Patient older than 65 years old, undergoing urgent abdominal surgery in our center
  Interventions: Procedure: surgery
- not surgical management: Patients that presents a surgical disease, but we desestimate surgical procedure

INTERVENTIONS:
Procedure: surgery
  Groups: surgical management

SUMMARY:
Morbimortality in older patients undergoing abdominal surgery.

DETAILED DESCRIPTION:
The aim of this study is to validate the modified CriSTAL tool for 30 mortality in elderly patients undergoing urgent abdominal surgery. To provide a new tool that could be used in conjunction with clinical judgment to aid in decision-making.

The second objective of our study was to assess the quality of life, frailty, functional status and nutritional status in elderly patients that survive six months after an urgent abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* >65 years old, accepted in emergency department

Exclusion Criteria:

* not sign the consent

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: patiens>65 years old
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Barthel index, questionnaire | 6 months
  to measure performance in activities of daily living

SECONDARY OUTCOMES:
Clavien- Dindo Modified | 1 year
  Morbimortality using Clavien-Dindo classification

OTHER OUTCOMES:
FRAIL scale, Fried score | 6 months
  To measure frailty

CONTACTS AND LOCATIONS:
Overall Officials: javier Herrera, doctor, Study Director — UPNA
Locations (1):
- UPNA, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No